CLINICAL TRIAL: NCT00473772
Title: Paclitaxel-Eluting PTCA-Balloon in Combination With the CoroflexTM Blue Stent vs the Sirolimus Coated CypherTM Stent in the Treatment of Advanced Coronary Artery Disease
Brief Title: DEBlue Stent vs Cypher Stent in the Treatment of Advanced Coronary Artery Disease
Acronym: PEPCADIII
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Collaborators: B.Braun Vascular Systems, Berlin, Germany (Unknown)
Responsible Party: Dr. Michael Boxberger, B.Braun Vascular Systems, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BBM-VS-54
Record Dates: First submitted 2007-05-14; First posted 2007-05-15 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Coronary Artery Disease
Keywords: cobalt chromium stent; paclitaxel coated balloon catheter; DEBlue; drug eluting balloon
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cypher Stent (Active Comparator)
  Interventions: Device: DEBlue stent vs. Cypher stent
- DEBlue Stent (Experimental)
  Interventions: Device: DEBlue stent vs. Cypher stent

INTERVENTIONS:
Device: DEBlue stent vs. Cypher stent — DES vs. DEB with BMS

SUMMARY:
The aim of the study is to assess the safety and efficacy of the Paclitaxel-eluting SeQuent Please S stent system (DEBlue) in the treatment of stenoses in native coronary arteries with nominal stent diameters between ≥ 2.5 mm and ≤ 3.5 mm and < 24 mm in length for procedural success and preservation of vessel patency in comparison to the Sirolimus-eluting CypherTM stent.

DETAILED DESCRIPTION:
The incidence of in-stent restenosis after percutaneous coronary intervention varies between 5 and 35% after bare metal stenting and is as high as 19% after the implantation of a drug-eluting stent in patients at moderate risk. Restenosis due to neointimal hyperplasia is a slow process, suggesting that therapeutic local drug administration would need to be prolonged to be beneficial. Stent-based local drug delivery provides sustained drug release using special release technologies like polymer coating. However, cell culture experiments indicate that even brief contact between vascular smooth muscle cells and lipophilic taxane compounds can inhibit vascular smooth muscle cell proliferation for a long period. In experiments in swine, intracoronary delivery of paclitaxel by contrast media or by a drug-coated balloon catheter was found to result in vascular tissue concentrations capable of producing antiproliferative effects, thus leading to a significant reduction in neointimal proliferation. In these animal studies, the most pronounced reduction of neointimal formation was seen with paclitaxel-coated balloon catheters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable or unstable angina or documented ischemia due to a significant lesion in a native coronary artery
* Patients eligible for coronary revascularization by means of PCI
* Intention to treat one lesion with one stent
* Patients suitable for coronary revascularization of any sort (balloon angioplasty, device-assisted balloon-angioplasty, or coronary artery bypass grafting)
* Patients must be ≥ 18 years of age
* Women of childbearing potential may not be pregnant nor have the desire to becoming pregnant during the first year following the study procedure. Hence, patients will be advised to use an adequate birth control method up to and including 9 months follow-up
* Patients who are mentally and linguistically able to understand the aim of the study and to show sufficient compliance in following the study protocol
* Patients must agree to undergo the 9 months angiographic follow-up
* Patients must agree to undergo the 1 and 3 year clinical follow-up
* Patient is able to verbally acknowledge an understanding of the associated risks, benefits, and treatment alternatives to therapeutic options of this trial, e.g. balloon angioplasty by means of the Paclitaxel-eluting PTCA-balloon catheter in combination with the Coroflex BlueTM stent or the Sirolimus-eluting CypherTM stent. The patients, by providing informed consent, agree to these risks and benefits as stated in the patient informed consent document.
* Significant stenoses in native coronary arteries with nominal stent diameters between ≥ 2.5 mm and ≤ 3.5 mm and < 24 mm in length

Exclusion Criteria:

* Unprotected left main
* In stent restenosis
* Indication for more than one lesion to treat, even as staged procedure
* Intended bifurcational stenting
* Patients requiring chronic anticoagulation
* SVG and AG
* Acute MI (STEMI, NSTEMI)
* Cardiogenic shock
* Chronic total occlusions
* Pregnancy
* Patients with stand alone balloon angioplasty, or stent deployment 6 months prior to enrolment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
late lumen loss | 9 months

SECONDARY OUTCOMES:
MACE | 9 months
MACE | 3 years
MACE | 30 days
Binary restenosis rate | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Scheller, Principal Investigator — University of Saarland - Internal Medicine III, Homburg/Saar, Germany; Christian Hamm, Principal Investigator — Kerckhoff-Clinic Bad Nauheim, Germany
Locations (16):
- Belgium (2):
  - Cardiovascular Center OLV Hospital Aalst, Aalst
  - Ziekenhuis Oost-Limburg, Genk
- Institute for Clinical and Experimental Medicine, Prague, Czechia
- Clinique Saint Martin, Caen, France
- Germany (8):
  - Klinik fuer Innere Medizin III, Universitaetsklinikum des Saarlandes, Homburg / Saar, Saarland
  - Kerckhoff-Clinic Bad Nauheim, Bad Nauheim
  - Kardiologie, Campus Virchow-Klinikum, Charite, Berlin
  - St. Johannes-Hospital, Dortmund
  - Medizinische Universitätsklinik III, Abt. Kardiologie und Angiologie, Freiburg im Breisgau
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Ludwigshafen, Ludwigshafen
  - University of Rostock, Rostock
- Rihnstate Hospital, Arnhem, Netherlands
- Hospital Universitari Germans Trias I Pujol, Badalona, Spain
- Universitetssjukhuset Lund, Lund, Sweden
- Northern General Hospital, Sheffield, United Kingdom

REFERENCES:
- [Background] Scheller B, Speck U, Bohm M. Prevention of restenosis: is angioplasty the answer? Heart. 2007 May;93(5):539-41. doi: 10.1136/hrt.2007.118059. PMID 17435062
- [Background] Scheller B, Hehrlein C, Bocksch W, Rutsch W, Haghi D, Dietz U, Bohm M, Speck U. Treatment of coronary in-stent restenosis with a paclitaxel-coated balloon catheter. N Engl J Med. 2006 Nov 16;355(20):2113-24. doi: 10.1056/NEJMoa061254. Epub 2006 Nov 13. PMID 17101615
- [Background] Speck U, Scheller B, Abramjuk C, Breitwieser C, Dobberstein J, Boehm M, Hamm B. Neointima inhibition: comparison of effectiveness of non-stent-based local drug delivery and a drug-eluting stent in porcine coronary arteries. Radiology. 2006 Aug;240(2):411-8. doi: 10.1148/radiol.2402051248. PMID 16864669
- [Background] Scheller B, Speck U, Abramjuk C, Bernhardt U, Bohm M, Nickenig G. Paclitaxel balloon coating, a novel method for prevention and therapy of restenosis. Circulation. 2004 Aug 17;110(7):810-4. doi: 10.1161/01.CIR.0000138929.71660.E0. Epub 2004 Aug 9. PMID 15302790
- [Background] Speck U, Scheller B, Abramjuk C, Bernhardt U. Drug delivery by angiographic contrast media: inhibition of restenosis. Acad Radiol. 2005 May;12 Suppl 1:S14-7. doi: 10.1016/j.acra.2005.02.017. No abstract available. PMID 16106539
- [Background] Speck U, Scheller B, Abramjuk C, Grossmann S, Mahnkopf D, Simon O. Inhibition of restenosis in stented porcine coronary arteries: uptake of Paclitaxel from angiographic contrast media. Invest Radiol. 2004 Mar;39(3):182-6. doi: 10.1097/01.rli.0000116125.96544.64. PMID 15076010
- [Background] Scheller B, Speck U, Schmitt A, Bohm M, Nickenig G. Addition of paclitaxel to contrast media prevents restenosis after coronary stent implantation. J Am Coll Cardiol. 2003 Oct 15;42(8):1415-20. doi: 10.1016/s0735-1097(03)01056-8. PMID 14563585
- [Background] Scheller B, Speck U, Romeike B, Schmitt A, Sovak M, Bohm M, Stoll HP. Contrast media as carriers for local drug delivery. Successful inhibition of neointimal proliferation in the porcine coronary stent model. Eur Heart J. 2003 Aug;24(15):1462-7. doi: 10.1016/s0195-668x(03)00317-8. PMID 12909076
- [Background] Scheller B, Speck U, Schmitt A, Clauss W, Sovak M, Bohm M, Stoll HP. Acute cardiac tolerance of current contrast media and the new taxane protaxel using iopromide as carrier during porcine coronary angiography and stenting. Invest Radiol. 2002 Jan;37(1):29-34. doi: 10.1097/00004424-200201000-00006. PMID 11753151